CLINICAL TRIAL: NCT06250452
Title: Effect of Halotherapy (Salt Therapy) on Oxygen Saturation (SPO2), Asthma Symptoms and Treatment Need in Children With Asthma
Brief Title: Effect of Halotherapy in Children With Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Igdir University (Other)
Responsible Party: Principal Investigator, Eda Gulbetekin, Assist. Prof., Igdir University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Eda1
Record Dates: First submitted 2024-01-23; First posted 2024-02-09 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Therapy, Oxygen Inhalation
Keywords: Halotherapy; Oxygen Saturation; Asthma; Children with Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): "Personal Information Form", SPO2 measurement and Asthma Symptom and Treatment Need Scoring / Daily Follow-up Form" will be applied to the children in the experimental group before they are taken to the salt therapy room.
  Interventions: Combination Product: Halotherapy (Salt Therapy)
- Control Group (Experimental): The same procedure will be applied to the children in the control group. In the study planned to be carried out for 6 weeks, it is recommended that children repeat the session for 10 minutes daily, the first 5 sessions every day and the other 5 weeks once a week.
  Interventions: Combination Product: Halotherapy (Salt Therapy)

INTERVENTIONS:
Combination Product: Halotherapy (Salt Therapy) — "Personal Information Form", SPO2 measurement and Asthma Symptom and Treatment Need Scoring / Daily Follow-up Form" will be applied to the children in the experimental group before they are taken to the salt therapy room. Scales and SPO2 measurement will be performed before, during and after therapy. The same procedure will be applied to the children in the control group, but no therapy will be applied. In the study planned to be carried out for 6 weeks, it is recommended that children repeat the session for 10 minutes daily, the first 5 sessions every day and the other 5 weeks once a week.

SUMMARY:
Introduction: Asthma is a chronic respiratory disease that can affect all age groups and is characterized by episodic and reversible wheezing, shortness of breath, chest tightness and cough attacks. According to a 2016 report by the United States Department of Disease Control and Prevention (CDC), the prevalence of asthma was 9.6% in children aged 5-11 and 10.5% in children aged 12-17. It has been shown that the prevalence of asthma under the age of 18, which concerns all childhoods, is 8.3%.

Purpose: The aim of the study is to determine the effect of salt therapy rooms on the oxygen saturation, asthma symptoms and treatment needs of children with asthma.

Material Method: The research was planned as an experimental study with experimental and control groups. Participants to be included in the study will be children between the ages of 4-10, diagnosed with asthma and without any other chronic diseases, who volunteer to participate. "Personal Information Form", "SPO2 measurements", "Asthma Symptom and Treatment Need Scoring / Daily Follow-up Form" and "Informed Voluntary Consent Form" will be used to collect data. The sample of the research was calculated using the GPower computer program. With power analysis, t-test in independent groups with a large effect size at α = 0.05 (d = 0.8) and in the calculation made to have a power of 95% of the study, it was found that a total of 70 children, 35 children in the control group and experimental groups, should be included. . "Personal Information Form", SPO2 measurement and Asthma Symptom and Treatment Need Scoring / Daily Follow-up Form" will be applied to the children in the experimental group before they are taken to the salt therapy room. The same procedure will be applied to the children in the control group. In the study planned to be carried out for 6 weeks, it is recommended that children repeat the session for 10 minutes daily, the first 5 sessions every day and the other 5 weeks once a week.

DETAILED DESCRIPTION:
"Salt therapy," known as halotherapy, is a treatment method performed in salt chambers lined with salt crystals that are pumped with salt-laden air and is used to combat respiratory diseases, skin conditions, mental fatigue and stress. The word Halos means salt in Greek. This practice is also performed in naturally occurring salt mines or caves in Eastern European countries, which is called "speleotherapy" or "cave salt therapy".

Salt has been used for thousands of years in different parts of the world due to its therapeutic effect, and was first applied for therapeutic purposes by Polish Feliks Bockowski. Although salt mine workers in Poland lack basic needs such as nutrition and have difficult working conditions, their general health has led researchers to study and observe in the salt field. In this observation, it was determined that mine workers were less likely to catch colds or any respiratory system diseases. Salt mines were thought to have health benefits, and salt caves in Eastern Europe and Poland became popular.

The research was planned as an experimental study with experimental and control groups. Participants to be included in the study will be children between the ages of 4-10, diagnosed with asthma and without any other chronic diseases, who volunteer to participate. "Personal Information Form", "SPO2 measurements", "Asthma Symptom and Treatment Need Scoring / Daily Follow-up Form" and "Informed Voluntary Consent Form" will be used to collect data. The sample of the research was calculated using the GPower computer program. With power analysis, t-test in independent groups with a large effect size at α = 0.05 (d = 0.8) and in the calculation made to have a power of 95% of the study, it was found that a total of 70 children, 35 children in the control group and experimental groups, should be included. . "Personal Information Form", SPO2 measurement and Asthma Symptom and Treatment Need Scoring / Daily Follow-up Form" will be applied to the children in the experimental group before they are taken to the salt therapy room. The same procedure will be applied to the children in the control group. In the study planned to be carried out for 6 weeks, it is recommended that children repeat the session for 10 minutes daily, the first 5 sessions every day and the other 5 weeks once a week.

ELIGIBILITY:
Inclusion Criteria:

* Asthma diagnosis
* Being a child between the ages of 4-10
* Volunteering to participate in research

Exclusion Criteria:

* Under 4 years of age and over 10 years of age
* Any other chronic disease
* not agree to participate in the research

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2024-03-06 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Oxygen Saturation (SPO2) | for 6 weeks, children were given 10-minute daily sessions, the first 5 sessions every day, the other 5 weeks, once a week.
  Oxygen saturation is a very important measure of how well the lungs are working.

SECONDARY OUTCOMES:
Asthma Symptom and Treatment Need Scoring | for 6 weeks, children were given 10-minute daily sessions, the first 5 sessions every day, the other 5 weeks, once a week.
  All patients were given a form to record their asthma symptoms at the beginning and end of the study. Daily symptoms (cough, wheezing, shortness of breath) were scored using the scoring system. In this scoring, symptom-free status was scored as 0, mild symptoms as 1, moderate symptoms as 2, and severe symptoms as 3.

CONTACTS AND LOCATIONS:
Overall Officials: Eda Gülbetekin, PhD, Principal Investigator — Igdir University
Locations (2):
- Turkey (Türkiye) (2):
  - Eda Gülbetekin, Iğdır, Iğdır
  - Eda Gülbetekin, Iğdır

IPD SHARING:
Plan to Share IPD: No